CLINICAL TRIAL: NCT00902850
Title: One-Day Dispensing Clinical Evaluation of SofLens Daily Disposable Lenses Compared to 1-Day Acuvue TruEye Lenses
Brief Title: One-Day Dispensing Clinical Evaluation of SofLens Daily Disposable Lenses Compared to a Marketed 1 Day Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ROC2-08-169
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Contact Lenses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SofLens Daily Disposable (Experimental): SofLens Daily Disposable Lenses
  Interventions: Device: SofLens Daily Disposable
- Marketed 1 Day Contact Lens (Active Comparator): Marketed 1 Day Contact Lens
  Interventions: Device: Marketed 1 Day Contact Lens

INTERVENTIONS:
Device: SofLens Daily Disposable — Lenses to be worn for 8-16 hours
  Arms: SofLens Daily Disposable
Device: Marketed 1 Day Contact Lens — Lenses to be worn for 8-16 hours
  Arms: Marketed 1 Day Contact Lens

SUMMARY:
The objective of this one-day study will be to evaluate the clinical performance of SofLens Daily Disposable lenses compared to that of a marketed 1 Day Contact Lens.

ELIGIBILITY:
Inclusion Criteria:

* Have physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings.
* Have no active ocular disease or allergic conjunctivitis.
* Not be using any topical ocular medications.

Exclusion Criteria:

* Participating in a conflicting study.
* Considered by the Investigator to not be a suitable candidate for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Steffen, OD, MS, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Research Clinic, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SofLens Daily Disposable | Marketed 1 Day Contact Lens
Started | 14 | 14
Completed | 12 | 12
Not Completed | 2 | 2
Not completed — Physician Decision | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SofLens Daily Disposable | Marketed 1 Day Contact Lens | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Median (Full Range); unit: years] | 40 [24 to 59] | 40 [24 to 59] | 40 [24 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Clinical Performance
Description: Comfort of lens wear compared at insertion of lens, 4 hours after insertion, and end of day (8-16 hours of wear-time). Score was a number on a scale 0-100, graded by the participants, and included lens edge awareness, scratchiness/grittiness, foreign body sensation, and general lens awareness.
Time Frame: Insertion, 4 hours & End of Day
Population: All eligible participants
Measure: Number; unit: units on a scale
Arm/Group | SofLens Daily Disposable | Marketed 1 Day Contact Lens
Number analyzed (Participants) | 12 | 12
units on a scale
  Lens Insertion | 98.1 | 100
  4 Hours after insertion | 97.5 | 98.1
  End of Day (8-16 hours) | 91.9 | 91.7

ADVERSE EVENTS:
Arm/Group | SofLens Daily Disposable | Marketed 1 Day Contact Lens
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes